CLINICAL TRIAL: NCT07236138
Title: The Interactive Distraction Technique for Controlling Gag Reflex During Endodontic Diagnostic Radiography of Posterior Teeth: A Split-Mouth Randomized Controlled Clinical Trial With Patients Reported Outcomes
Brief Title: Controlling Gag Reflex During Endodontic Diagnostic Radiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Muhammad Zubair Ahmad, Associate Professor, Qassim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-14-11
Record Dates: First submitted 2025-04-23; First posted 2025-11-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gagging; Satisfaction, Patient; Endodontic Disease; Anxiety; Xray Complication
Keywords: distraction; endodontic diagnosis; gag reflex; periapical radiograph; virtual reality
MeSH Terms: conditions — Gagging; Patient Satisfaction; Dental Pulp Diseases; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized split-mouth (within-subject) parallel design. This was a randomized split-mouth clinical trial in which the intervention and control were allocated to two different sides of the mouth within the same participant. Allocation of the intervention side was determined by randomization. Both interventions were delivered during the same visit, with no time-based sequence or washout period. Each participant therefore served as their own control, receiving both the intervention and control concurrently at different intra-oral sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1. Periapical radiograph without virtual reality (VR) distraction (Other): In this group an experienced endodontist will take Digital periapical radiographs using photostimulable phosphor plates (DigoraOptime, Soredex Medical Systems, Helsinki, Finland), with a holder for standardization and a paralleling technique for ortho-radial projection at a focus-receptor distance of 20 cm. The size of the plates will be selected according to the patient's arch size. Plates will be exposed using a De Gotzen X-Mind® Unity X-ray unit (De Gotzen Srl, Olgiate Olona, Italy), set at 70 kVp and 8 mA, with an exposure time of 0.25 seconds. The radiograph will be taken.
  Interventions: Other: Periapical radiograph will be taken without VR
- Group 2. Periapical radiograph with virtual reality (VR) distraction (Experimental): In this group all steps will remain the same as comparator group except that periapical radiograph will be taken using following virtual reality (VR) distraction approach.
  An Oculus Quest VR headset will be used in this study. Each participant will be briefly instructed regarding the interactive distraction VR device. The VR headset will be loaded with a short, animated movie, which will be shown to each participant in the experimental group (G2) two minutes before the procedure. Each patient will fill out a modified dental anxiety scale prior to radiography procedures.
  Interventions: Device: Periapical radiograph will be taken with VR

INTERVENTIONS:
Other: Periapical radiograph will be taken without VR — In the comparison group no intervention will be used. Standard periapical radiographs will be taken for endodontic diagnostic procedure.
  Arms: Group 1. Periapical radiograph without virtual reality (VR) distraction
Device: Periapical radiograph will be taken with VR — The VR headset will be loaded with a short, animated movie, which will be shown to each participant in the experimental group two minutes during the standard periapical radiographs taking procedure.
  Arms: Group 2. Periapical radiograph with virtual reality (VR) distraction

SUMMARY:
Intraoral radiography plays a vital role in endodontic diagnosis and treatment planning. However, many patients experience discomfort during periapical radiographic procedures due to factors such as a pronounced gag reflex and dental anxiety, making the process difficult and distressing. Managing these issues is essential for enhancing patient cooperation and improving overall treatment experience.

This study investigates the potential of Virtual Reality (VR) interactive distraction as a noninvasive method to control gag reflex and improve patient comfort during intraoral radiography. While VR has shown promise in reducing dental anxiety in various procedures, its effectiveness in managing gag reflex during diagnostic endodontic radiography remains largely unexplored.

The primary objective of this study is to evaluate the effectiveness of VR in reducing the gag reflex in adult patients undergoing routine periapical radiographs for maxillary molar teeth. Secondary objectives include assessing patient preferences, experiences, and satisfaction associated with the use of VR.

The study involves patients who require bilateral intraoral diagnostic radiographs of maxillary molars. Each patient will undergo two radiographs: one with standard procedure (Control - Group 1), and the other using VR distraction (Experimental - Group 2). A randomized, computer-generated list will determine which side will receive the VR intervention.

Gag reflex scores will be measured before and after the procedure, pre- and post-procedure anxiety levels will be recorded using Modified Dental Anxiety Scale (MDAS). Additionally, a structured questionnaire will assess patient satisfaction and experience with the VR device. Physiological indicators such as pulse rate, blood pressure, and oxygen saturation will be recorded to evaluate any changes associated with the use of VR.

This study aims to generate evidence on whether VR distraction can be an effective tool for controlling gag reflex and improving patient tolerance, ultimately enhancing the quality of care in diagnostic dental radiography.

DETAILED DESCRIPTION:
Background:

Intraoral radiography is crucial for accurate endodontic diagnosis and treatment planning. However, some patients face challenges during periapical radiography procedures. Many struggle to tolerate the placement of intraoral films or sensors; a problem worsens because of gag reflexes and dental anxiety.

Rationale:

Controlling gag reflexes, improving patient experience, and reducing anxiety are priorities in all dental procedures. Virtual reality (VR) interactive distraction is a promising noninvasive tool to improve patient experience and reduce anxiety during dental procedures. So far, little to no evidence exists regarding the impact of VR on controlling gag reflex in patients undergoing diagnostic endodontic intraoral radiography procedures.

Study objectives:

As its primary objective, this study will evaluate the use of VR interactive distraction to control the gag reflex in adult patients undergoing routine endodontic diagnostic intraoral radiography for maxillary molar teeth. As its secondary objectives, the study will evaluate the impact of VR on patients' preferences, experiences, and satisfaction as well as anxiety levels.

Methods:

The study will be conducted on patients who require endodontic bilateral diagnostic intraoral radiographs of maxillary molar teeth for reasons not related to this study. Two radiographs will be taken for each patient as follows.

* Control (G1) - Periapical radiograph without application of VR distraction.
* Experimental (G2) - Periapical radiograph with the application of VR distraction.

A computer-generated list will be used to randomly select the control and experimental sides. Modified Dental Anxiety Scale (MDAS) will be used to assess anxiety before and after finishing the radiography procedures. A structured questionnaire will be used to evaluate the satisfaction and experience regarding using a Virtual reality device. The pulse rate, blood pressure, and oxygen saturation will be measured for physiological assessment at three timepoints (pre-procedure, during procedure and post-procedure).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old) visiting the Al-Rass dental clinics of the College of Dentistry and undergoing bilateral maxillary molar periapical radiographs for endodontic diagnostic purposes.
* Patients who are willing to collaborate in the study and willing to sign the written informed consent.
* Classified as class I, II according to the American Society of Anesthesiologists Physical Status Classification System.
* Patients exhibiting a gag reflex of "moderate" to "very severe" according to the classification of the Gagging Problem (CGP) index

Exclusion Criteria:

* Mentally or medically compromised patients.
* Patients with acute pain, such as acute pulpitis, which require emergency treatment.
* Pregnant women.
* Patients on any medications for the past two weeks.
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Severity of gagging | Baseline (pre-procedure) and periprocedural (during X-ray film placement) on Day 1.
  The 5-point Gagging Severity (GS) Scale will be used to assess the change in gagging response between the two study arms. In this scale, G1 = no gagging and G5 = very severe gagging; higher scores indicate a worse gag reflex.

SECONDARY OUTCOMES:
Dental anxiety | Immediately before and immediately after the radiographic procedure (Day 1).
  Dental anxiety will be assessed using the 5-item Modified Dental Anxiety Scale (MDAS). Each item is scored from 1 (not anxious) to 5 (extremely anxious), with a total score range of 5-25; higher scores indicate greater anxiety.
Physiological response (pulse rate, blood pressure, and oxygen saturation) | Before, during, and after the radiographic procedure (Day 1).
  Physiological parameters, including pulse rate (beats per minute), blood pressure (mmHg), and oxygen saturation (%), will be recorded to evaluate physiologic changes during virtual reality distraction.
Patient preferences, experiences, and satisfaction | Immediately after X-ray film placement (post-procedural, Day 1).
  A structured questionnaire using a 5-point Likert scale will be used to evaluate patients' preferences, experiences, and satisfaction with the virtual reality device during intraoral radiography.
  Each item is scored from 1 (very dissatisfied / strongly disagree) to 5 (very satisfied / strongly agree); higher scores indicate a more favorable experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Muhammad Zubair Ahmad, Ar Rass, Al-Qassim Region, Saudi Arabia